CLINICAL TRIAL: NCT02248948
Title: Multicenter Randomized Controlled Trial for the Evaluation of Superiority of a Supplement With Omega-3 Fatty Acids Versus Placebo for the Improvement of Attention Deficit and Hyperactivity Disorder (ADHD) in Children
Brief Title: Superiority of Omega-3 Versus Placebo on the Improvement of ADHD in Children
Acronym: ECOMEGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratorios Ordesa (Industry)
Collaborators: Clever Instruments S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ECOMEGA-TDAH-014; 2013-004638-14 (EudraCT Number)
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: Omega-3; ADHD; Quality of Life; Inattention; Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medium Chain Triglycerides Supplement (Placebo Comparator): Medium Chain Triglycerides Oil with 5 micrograms of Vitamin D and 6 mg of Vitamin E in 4 ml.
  Interventions: Dietary Supplement: Medium Chain Triglycerides
- Omega-3 Fatty Acids Supplement (Experimental): The Omega-3 Fatty Acid supplement provides 540 mg of eicosapentaenoic acid (EPA), 340 mg of docosahexaenoic acid (DHA), 60 mg of gamma linolenic acid (GLA/Omega-6), 5 micrograms of Vitamin D and 6 mg of Vitamin E in 4 ml.
  Interventions: Dietary Supplement: Omega-3 Fatty Acids

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acids — Patients will receive a daily dose calculated based on the child weight (≤28 kg=4ml; 29-40 kg= 6ml and ≥41 kg=8ml) and will be provided once a day for 6 months.
  Other Names: EPA/DHA
  Arms: Omega-3 Fatty Acids Supplement
Dietary Supplement: Medium Chain Triglycerides — Patients will receive a daily dose calculated based on the child weight (≤28 kg=4ml; 29-40 kg= 6ml and ≥41 kg=8ml) and will be provided once a day for 6 months.
  Other Names: Placebo
  Arms: Medium Chain Triglycerides Supplement

SUMMARY:
This study aims to evaluate the efficacy of an Omega-3 Fatty Acid Supplement on improving the Attention Deficit Hyperactivity Disorder (ADHD) clinical symptoms.

DETAILED DESCRIPTION:
This is a multicenter, controlled, randomized, prospective, parallel-group, double-blind study to evaluate the effect of an Omega-3 Fatty Acid Supplement with EPA, DHA, vitamins E and D on ADHD clinical symptoms (according to Diagnostic and Statistical Manual for Mental Disorders, 4th. edition (DSM-IV-TR) criteria) in children between 6 and 11 years. Patients will be randomized to receive either the new omega-3 supplement or a placebo during 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 11 years 11 months.
* ADHD diagnosis according to DSM-IV-TR criteria
* Children whose parents are able to reliably meet all visits and all the tests required for this study based on the researcher judgment
* Patient representative (either parents or legal guardians) must understand the conditions of the study and sign the informed consent

Exclusion Criteria:

* Patients who do not meet diagnostic criteria for ADHD
* Patients with a previously known allergy or intolerance to the components of Omega- 3 supplement
* Patients with underlying diseases that, according to medical criteria , are not eligible for supplementation with Omega-3 fatty acids : fatty liver disease (or other liver disease), bleeding disorders and cardiovascular disease
* Patients with allergies to fish and /or shellfish
* Patients who have received ADHD pharmacological treatment or fatty acid supplements at any dose for more than 7 consecutive days within the last 3 months
* Patients who have received psychological or psycho-educational treatment in the past 3 months
* Patients who have had some kind of psychometric diagnostic tests in the last year
* Patients with scores corresponding to a lower mental age (more than 1 year less) according to the Wechsler Intelligence Cubes Scale for Children (WISC-IV)
* Patients with severe emotional problems according to the CAS or STAIC tests
* Patients participating in another clinical trial

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 231 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Improvement in clinical symptoms of ADHD | At baseline and at 6 months
  Differences between groups measured by:
  1. Number of criteria of the ADHD-Scale-IV rated by parents and teachers
  2. Clinical Global Impressions Scale (CGI) assessed by the physician

SECONDARY OUTCOMES:
Changes in neuropsychological outcomes | At baseline and at 6 months
  Differences between groups measured by Scores of the Conners Continuous Performance Test-II (CPT-II) which evaluate potential problems related to executive functions perception, internal ordering, working memory, motor control.
Changes in emotional outcomes | At baseline and at 6 months
  Differences between groups measured by Cognitive Assessment System (CAS) for children between 6-8 years old and by State-Trait Anxiety Inventory for Children (STAIC) for children between 9-12 years old.
Changes in Children's Quality of Life | At baseline and at 6 months
  Differences between groups measured with Child Health and Illness Profile- Parent Form (CHIP-CE)
Changes in Quality of Life of Parents of Children with ADHD | At baseline and at 6 months
  Differences between groups measured with a Short Version of the World Health Organization Quality of Life Instruments (WHOQoL)

OTHER OUTCOMES:
Changes in nutritional status | At baseline and at 2, 4 and 6 months
  Differences between groups measured by anthropometry and feeding scale of the Health National Survey (National Statistical Institute, Spain).
Tolerability of study product | At 2, 4 and 6 months
  Differences between groups measured by product acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Sasot Llevadot, MD, Principal Investigator — Centro Médico Teknon; Ana Bielsa, MD, Study Chair — Unidad Clínica Familianova Schola; Miquel Sisteré, MD, Study Chair — Centre de Salut Mental Infanto-Juvenil, Lleida; Esther Cardo Jalón, MD, Study Chair — Unidad Pediártica Balear, Palma de Mallorca; Isabel Hernández Otero, MD, Study Chair — Hospital Universitario Virgen de la Victoria, Málaga.
Locations (1):
- Centro Médico Teknon, Barcelona, Spain

REFERENCES:
- [Derived] Gillies D, Leach MJ, Perez Algorta G. Polyunsaturated fatty acids (PUFA) for attention deficit hyperactivity disorder (ADHD) in children and adolescents. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD007986. doi: 10.1002/14651858.CD007986.pub3. PMID 37058600